CLINICAL TRIAL: NCT04339686
Title: Multicentric Retrospective Observational Study of Thoracic Scanner Performance in COVID Screening. Comparison to Virological Testing and Multiparametric Gold Standard
Brief Title: Multicentric Retrospective Observational Study of Thoracic Scanner Performance in COVID Screening.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: POWER-COVID_CT
Record Dates: First submitted 2020-04-08; First posted 2020-04-09 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: The Gold Standard for Current SARS CoV2 Detection is RT-PCR

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Suspicion of COVID 19
  Interventions: Diagnostic Test: Thoracic CT Scan

INTERVENTIONS:
Diagnostic Test: Thoracic CT Scan — Retrospective analysis of the thoracic CT scan results compared to final discharge summary

SUMMARY:
All patients included in this search will be on anonymized file: Symptomatic patients consulting for suspicion of COVID 19 with indication to a screening (RT-PCR, Scanner) according to the criteria of the Ministry of Health.

To evaluate the diagnostic performance of chest CT in screening for COVID-related lung injury in patients with a clinical suspicion of COVID.

CT scan results for COVID according to French thoracic imaging society will be dichotomized into evocative or compatible (considered positive) non-evocative (considered negative) The results will be compared to the gold standard corresponding to a multiparametric element: the discharge summary.

Ct Scan performance will be recorded and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* All patients suspected of COVID 19 consulting for diagnostic

Exclusion Criteria:

* Delay between RT-PCR and Thoracic Scan greater than 6 days.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients suspected of COVID 19 consulting for diagnostic
Sampling Method: Non-Probability Sample
Enrollment: 56000 (Estimated)
Dates: Start 2020-04-20 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of chest CT in screening for pulmonary lesions in clinical suspicions of COVID. | 1 month
  CT Report will dichotomized into evocative or non-evocative for COVID-related lung injury.

SECONDARY OUTCOMES:
Compare the diagnostic performance of chest CT and RT-PCR in COVID 19 at the initial consultation (screening). | 1 month
  Initial virological RT-PCR results: positive or negative depending on the laboratories of the institutions.
  Scanner results according to French Thoracic Imaging Society.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: No